CLINICAL TRIAL: NCT01587924
Title: A Four-week, Phase IIa, Randomized, Active-controlled, Parallel-group, Multi-center Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Switching Subjects From a Stable Dose of Recombinant Human Erythropoietin to GSK1278863 in Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease
Brief Title: 4 Week Switch Study in Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 116582
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-08

CONDITIONS: Anaemia
Keywords: Renal Impairment; Anemia; pharmacokinetics; hemodialysis; Chronic kidney disease; GSK1278863; hemoglobin; Prolyl hydroxylase inhibitor; recombinant human erythropoietin; erythropoiesis stimulating agents; Dialysis, Renal
MeSH Terms: conditions — Anemia; Renal Insufficiency; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.5 mg GSK1278863 (Experimental): once daily
  Interventions: Drug: GSK1278863
- 2 mg GSK1278863 (Experimental): once daily
  Interventions: Drug: GSK1278863
- 5 mg GSK1278863 (Experimental): once daily
  Interventions: Drug: GSK1278863
- rhEPO (Active Comparator): as required
  Interventions: Drug: rhEPO

INTERVENTIONS:
Drug: GSK1278863 — tablet
  Arms: 0.5 mg GSK1278863; 2 mg GSK1278863; 5 mg GSK1278863
Drug: rhEPO — injection
  Arms: rhEPO

SUMMARY:
This is a four-week, Phase IIa, randomized, active-controlled, parallel-group, multi-center study to evaluate the safety, efficacy and pharmacokinetics of switching subjects from stable rhEPO to GSK1278863 in approximately 68 hemodialysis-dependent subjects with anemia associated with chronic kidney disease. The study consists of a screening phase of 2 weeks, a 4-week treatment phase and a 2-week follow-up phase. The range of Hgb values for study eligibility is 9.5-12.0 g/dL and the subjects must have received the same rhEPO product with total weekly doses that varied by no more than 50% during the 4 weeks prior to the Screening visit (Week -1. This study aims to estimate the relationship between dose of GSK1278863 and Hgb response in hemodialysis-dependent (HDD) subjects with anemia associated with chronic kidney disease after switching from a stable maintenance dose of recombinant human erythropoetin (rhEPO).

DETAILED DESCRIPTION:
This is a four-week, Phase IIa, randomized, active-controlled, parallel-group, multi-center study to evaluate the safety, efficacy and pharmacokinetics of switching subjects from stable rhEPO to GSK1278863 in approximately 68 hemodialysis-dependent subjects with anemia associated with chronic kidney disease. The study consists of a screening phase of 2 weeks, a 4-week treatment phase and a 2-week follow-up phase. The range of Hgb values for study eligibility is 9.5-12.0 g/dL and the subjects must have received the same rhEPO product with total weekly doses that varied by no more than 50% during the 4 weeks prior to the Screening visit (Week -1. Eligible subjects, stratified by their prior rhEPO dose will be randomized in equal proportions to receive double-blind GSK1278863 0.5 mg, 2 mg or 5 mg QD (after discontinuing their rhEPO), or to continue to receive their existing type and dose of rhEPO (epoetins or their biosimilars, or darbepoetin). Study treatment will be stopped if Hgb values fall outside of the protocol pre-specified ranges. Subject completion is defined as completion of all study phases including the follow-up phase.

This study aims to estimate the relationship between dose of GSK1278863 and Hgb response in hemodialysis-dependent (HDD) subjects with anemia associated with chronic kidney disease after switching from a stable maintenance dose of recombinant human erythropoetin (rhEPO). In addition, the study will characterize the effect of GSK1278863 on various pharmacokinetic (PK)/pharmacodynamic (PD) markers, and will investigate the safety and tolerability of GSK1278863.

An early interim analysis of the Hgb data is planned after approximately 20 subjects from cohort 1 have completed 3 weeks of treatment. Depending upon the interim findings, a second cohort of subjects may be added to investigate an additional GSK1278863 dose arm. Recruitment to the first cohort will continue during the interim analysis.

A second interim analysis is planned after approximately 48 subjects from cohort 1 have completed 4 weeks treatment. The purpose of this interim is three-fold, to investigate if a second cohort of subjects may be added, to facilitate early development of dose-response and PK/PD statistical models, and to generate interim results to facilitate design and dosing decisions for the next trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age and weight: >/=18 years of age and >/=45 kg (weight post-dialysis).
2. On three times weekly hemodialysis for at least 8 weeks, irrespective of eGFR values and stage of chronic kidney disease (CKD).
3. A single-pool Kt/Vurea of >/=1.2 based on a historical value obtained within the prior month in order to ensure the adequacy of dialysis. If Kt/Vurea is not available, then an average of the last 2 values of urea reduction ratio (URR) of at least 65%.
4. rhEPO use: Using the same rhEPO (epoetins or darbepoetin) with total weekly doses that varied by no more than 50% during the prior 4 weeks (i.e., maximum vs. minimum total weekly doses </=50%).
5. Hgb concentrations 9.5-12.0 g/dL (inclusive).
6. Vitamin B12 above the lower limit of the reference range (may rescreen in two months).
7. Folate: >/= 2.0 ng/mL (may rescreen in one month).
8. Ferritin: >/=40 ng/mL with the absence of microcytic or hypochromic RBCs.
9. Transferrin saturation (TSAT): Within the reference range.
10. Iron replacement therapy: Stable maintenance dose of oral iron replacement therapy, if required, that will be maintained throughout the study. NOTE: IV iron replacement therapy is not allowed the two weeks prior to Screening through the end of the study (Week 6).
11. QTc: QTcB <470 msec or QTcB <480 msec in subjects with bundle branch block obtained at Screening Visit (based on Central Reader's interpretation).
12. Females: Eligible to participate if she is of childbearing potential, and must agree to use one of the approved contraception methods from Screening until completion of the Follow-up Visit OR of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation of hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH)>40MIU/ml and estradiol <40pg/ml is confirmatory]. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
13. Males: Must agree to use one of the approved contraceptive methods from the time of Screening until completion of the Follow-up Visit.

Exclusion Criteria:

1. Dialysis modality: On peritoneal dialysis OR planned change in dialysis modality within the study time period.
2. rhEPO Hyporesponders: As defined by an epoetin dose of >/=360 IU/kg/week IV or darbepoetin dose of >/=1.8 µg/kg/week IV within the prior 8 weeks.
3. Renal transplant: Renal transplant anticipated or scheduled within the study time period or subjects with a functioning renal transplant.
4. Mircera or Peginesatide: Current or prior use (within the prior 8 weeks) of Mircera (methoxy polyethylene glycol epoetin beta) OR peginesatide.
5. Total CPK: >5x the upper limit of the reference range.
6. HIV: Positive HIV antibody.
7. History of myocardial infarction or acute coronary syndrome within the prior 6 months.
8. History of stroke or transient ischemic attacks (TIAs) within the prior 6 months.
9. Heart failure: Class III/IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
10. Hypertension: Poorly controlled hypertension, whether due to inadequate treatment, or lack of treatment, is defined as follows:

    * DBP >100 mmHg or SBP>160 mmHg for subjects taking hypertension medication(s) before screening and dialysis, if required.
    * DBP >105 mmHg or SBP>170 mmHg for subjects who are asked to hold hypertension medication(s) before screening and dialysis.
11. Thrombotic Disease: History of thrombotic disease (e.g., venous thrombosis such as deep vein thrombosis or pulmonary embolism, or arterial thrombosis such as new onset or worsening limb ischemia requiring intervention), or other thrombosis related condition except shunt thrombosis) within the prior 6 months.
12. Pulmonary hypertension: Known pulmonary hypertension and those at higher risk (than normally associated with CKD) for pre-existing elevation in pulmonary pressure (e.g., significant heart failure or lung disease requiring supplemental oxygen, or those with connective tissue diseases).
13. Inflammatory disease: Chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease).
14. Haematological disease: Any haematological disease including those affecting platelets, the coagulation disorders (e.g., Protein C or S deficiency) or red blood cells (e.g. sickle cell anemia, myelodysplastic syndromes, haematological malignancy, myeloma, haemolytic anemia) or any other cause of anemia other than renal disease.
15. Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alkaline phosphatase, alanine transaminase (ALT) or aspartate transaminase (AST) > 2.0 x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN]; or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participation in the study.
16. Major surgery: (excluding vascular access surgery) Within the prior 12 weeks or planned during the study.
17. Transfusion: Blood transfusion within the prior 12 weeks or an anticipated need for blood transfusion during the study.
18. Ulcer and Active GI Bleeding: Evidence of active peptic, duodenal, or esophageal ulcer disease OR GI bleeding within the prior 12 weeks.
19. Acute infection: Clinical evidence of acute infection or history of infection requiring intravenous (IV) antibiotic therapy the eight weeks prior to Screening through Day 1 (randomization).
20. Malignancy: History of malignancy within the prior 5 years or are receiving treatment for cancer or those with a strong family history of cancer (e.g., familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated.
21. Eyes: History of proliferative retinopathy requiring treatment within the prior 12 months or macular edema requiring treatment.
22. Severe reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
23. Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from Screening until the Follow-up Visit.
24. Androgens: New androgen therapy or changes to pre-existing androgen regimen within the prior 12 weeks.
25. Prior investigational product exposure: The Subject has participated in a clinical trial and has received an experimental investigational product within the prior 30 days.
26. Protocol compliance: Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
27. Other Conditions: Any condition which in the investigator's opinion should exclude the subject from participating in the study.
28. Pregnancy or Lactation: Pregnant females as determined by positive serum hCG test OR women who are lactating at Screening or during the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05-23 (Actual); Primary Completion 2013-05-27 (Actual); Study Completion 2013-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (56):
- United States (37):
  - GSK Investigational Site, Paragould, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Pine Bluff, Arkansas
  - GSK Investigational Site, Azusa, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Lynwood, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Arvada, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Westminster, Colorado
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Spring Hill, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Southgate, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Greenville, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, San Antonio, Texas
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
- Denmark (3):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Odense
  - GSK Investigational Site, Roskilde
- Germany (7):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Oberschleißheim, Bavaria
  - GSK Investigational Site, Lehrte, Lower Saxony
  - GSK Investigational Site, Demmin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Oslo, Norway
- Sweden (3):
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Holdstock L, Meadowcroft AM, Maier R, Johnson BM, Jones D, Rastogi A, Zeig S, Lepore JJ, Cobitz AR. Four-Week Studies of Oral Hypoxia-Inducible Factor-Prolyl Hydroxylase Inhibitor GSK1278863 for Treatment of Anemia. J Am Soc Nephrol. 2016 Apr;27(4):1234-44. doi: 10.1681/ASN.2014111139. Epub 2015 Oct 22. PMID 26494831
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in hemodialysis-dependent (HDD) participants from 06 June 2012 till 17 June 2013 across 48 centers in the United States (US), Canada, and European Union. A total of 68 participants were planned to be enrolled.
Pre-assignment Details: A total of 103 participants were screened, out of which 83 participants were randomized in the study. The participants were receiving recombinant human erythropoietin (rhEPO) for 2 weeks and had hemoglobin (hgb) range of 9.5 to 12.0 gram per deciliter (g/dL); however, one participant did not receive the study drug.
Groups:
- 0.5 mg GSK1278863: Eligible participants received oral GK1278863 0.5 milligrams (mg) once daily for 4 weeks and we re followed-up for 2 weeks
- 2 mg GSK1278863: Eligible participants received oral GK1278863 2.0 mg once daily for 4 weeks and were followed-up for 2 weeks
- 5 mg GSK1278863: Eligible participants received oral GK1278863 5.0 mg once daily for 4 weeks and were followed-up for 2 weeks.
- rhEPO: Eligible participants received oral rhEPO or darbepoetin once daily for 4 weeks and were followed-up for 2 weeks
Period: Overall Study
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Started | 21 | 21 | 21 | 20
Completed | 17 | 17 | 17 | 19
Not Completed | 4 | 4 | 4 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 2 | 1
Not completed — Met Hemoglobin stopping criteria | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included all randomized participants who received at least one dose of the study drug, had a baseline and at least one corresponding on treatment laboratory assessment.
Groups:
- 0.5 mg GSK1278863: Eligible participants received oral GK1278863 0.5 mg once daily for 4 weeks and we re followed-up for 2 weeks
- Total: Total of all reporting groups
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO | Total
Number analyzed (Participants) | 21 | 20 | 19 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (16.80) | 54.7 (18.78) | 55.9 (18.37) | 64.2 (12.77) | 57.8 (16.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 8 | 4 | 22
  Male | 18 | 13 | 11 | 16 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 4 | 4 | 18
  White | 14 | 14 | 12 | 14 | 54
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Modeled Hemoglobin (Hgb) Change From Baseline (Pre-dose on Day 1) at 4 Weeks of Treatment
Description: Modeled Hgb change from Baseline over 4 weeks of treatment. Change from Baseline is the actual value of Hgb at Week 4 minus the Baseline value. For modeled change at Week 4 participants required a Baseline and two or more non missing post-baseline values. Baseline is the average of Week -2, -1 and Day 1 values. The model included fixed effects for Baseline Hgb, treatment, and treatment by day interaction. Covariate analysis for modeled Hgb change was performed. Random effects were fitted in the intercept and the slope over time.
Time Frame: Baseline (pre-dose on Day 1) and up to week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 20 | 20 | 18 | 19
Grams per deciliter (g/dL) | -1.130 (0.6830) | -1.070 (0.7703) | 0.212 (0.7521) | -0.273 (0.6335)
Statistical Analysis 1: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline Hgb <10.80 versus modeled Hgb change from baseline in participants with Baseline Hgb >= 10.80; Test type: Superiority or Other; p = 0.0135, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 2: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline weight <= 80.5 Kg versus modeled Hgb change from baseline in participants with Baseline weight > 80.5; Test type: Superiority or Other; p = 0.5082, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 3: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with ethnicity non-Hispanic or Latino versus modeled Hgb change from baseline in participants with ethnicity non-Hispanic or Latino; Test type: Superiority or Other; p = 0.9770, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 4: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline geographic ancestry as African American versus modeled Hgb change from baseline in participants with no geographic ancestry as African American; Test type: Superiority or Other; p = 0.0618, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 5: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline gender as male versus modeled Hgb change from baseline in participants with Baseline gender female; Test type: Superiority or Other; p = 0.7495, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 6: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline age <65 years versus modeled Hgb change from baseline in participants with Baseline age >=65 years; Test type: Superiority or Other; p = 0.7865, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 7: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline co-ad with food versus modeled Hgb change from baseline in participants with Baseline co-ad without food; Test type: Superiority or Other; p = 0.0622, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 8: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline diabetes presence versus modeled Hgb change from baseline in participants with no Baseline diabetes; Test type: Superiority or Other; p = 0.2044, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day
Statistical Analysis 9: Comparison: 0.5 mg GSK1278863 vs 2 mg GSK1278863 vs 5 mg GSK1278863 vs rhEPO; Modeled Hgb change from baseline in participants with Baseline region as the US and Canada versus modeled Hgb change from baseline in participants with Baseline region as not the US and Canada; Test type: Superiority or Other; p = 0.8537, Regression, Linear — The p-value is showing the interaction of each subgroup by treatment and by day

2. Secondary Outcome: Hgb Variability Over 4 Weeks
Description: Within participant standard deviation for Hgb acts as a measure of Hgb variability. Hgb of participants was recorded over 4 weeks.
Time Frame: Up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 20 | 20 | 18 | 19
g/dL | 0.53 (0.271) | 0.55 (0.325) | 0.40 (0.364) | 0.35 (0.193)

3. Secondary Outcome: Evaluation of Change From Baseline in Hepcidin Over Period
Description: Evaluation of change from baseline for hepcidin was performed over 4 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was the last pre-dose value. Adjusted mean change from Baseline is presented as Least square (LS) mean.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Micrograms per liter (mcg/L)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 18 | 17 | 17 | 18
Micrograms per liter (mcg/L) | 204.88 (60.741) | 150.29 (62.619) | 16.42 (62.815) | -45.47 (61.939)

4. Secondary Outcome: Evaluation of Change From Baseline (Pre-dose on Day 1) in High Sensitivity C-Reactive Protein (hsCRP) Over 4 Weeks
Description: Evaluation of change from Baseline for hsCRP was analyzed over 4 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was the last pre-dose value. Peak change from Baseline also was calculated; however adjusted mean change from Baseline has been presented here as LS means.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Milligrams per liter (mg/L)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 19 | 18 | 17 | 19
Milligrams per liter (mg/L) | -0.40 (1.784) | -4.76 (1.834) | -1.48 (1.886) | -2.92 (1.784)

5. Secondary Outcome: Change From Baseline for Erythropoeitin (EPO) Over Period
Description: Evaluation of change from Baseline (pre-dose on Day 1) for EPO was analyzed over 4 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was the pre-dose Day 1 value. Adjusted means are presented as LS means.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Units per liter (U/L)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 18 | 18 | 16 | 19
Units per liter (U/L) | 4.368 (73.3485) | 3.263 (73.5023) | 181.948 (77.7763) | 393.159 (71.4855)

6. Secondary Outcome: Evaluation of Change From Baseline (Pre-dose on Day 1) for Peak Vascular Endothelial Growth Factor (VEGF) Over 4 Weeks
Description: Evaluation of change from Baseline for peak VEGF was analyzed up to 4 weeks. Baseline assessment was performed pre-dose on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Absolute mean change and peak change from Baseline in peak VGEF were also calculated; however, only model adjusted peak change in peak VGEF from Baseline has been presented as LS means.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms per liter (ng/L)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 19 | 18 | 17 | 17
Nanograms per liter (ng/L) | 23.21 (12.110) | 21.52 (12.291) | 53.85 (12.645) | 20.59 (12.874)

7. Secondary Outcome: Evaluation of Change From Baseline (Pre-dose on Day 1) for Hematocrit Over 4 Weeks
Description: Evaluation of change from Baseline for hematocrit over 4 weeks was performed. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 20 | 19 | 20
Percentage
  Week 1: number analyzed (Participants) | 19 | 20 | 19 | 18
  Week 1 | -0.59 (1.609) | -0.16 (1.823) | -0.75 (1.735) | 0.20 (1.738)
  Week 2: number analyzed (Participants) | 19 | 20 | 17 | 19
  Week 2 | -1.33 (2.122) | -1.56 (2.296) | -0.75 (1.960) | 2.02 (8.248)
  Week 3: number analyzed (Participants) | 16 | 17 | 17 | 18
  Week 3 | -2.32 (2.634) | -2.22 (2.712) | -0.65 (2.277) | 0.24 (2.507)
  Week 4: number analyzed (Participants) | 18 | 18 | 15 | 19
  Week 4 | -3.22 (2.731) | -2.63 (3.006) | -0.33 (2.044) | -0.22 (2.874)

8. Secondary Outcome: Residual Standard Deviation in Hgb (From the Linear Regression)
Description: Residual standard deviation was derived by linear regression. Hgb of participants was recorded over 4 weeks
Time Frame: Up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 20 | 20 | 18 | 19
g/L | 0.24 (0.108) | 0.26 (0.115) | 0.26 (0.309) | 0.20 (0.112)

9. Secondary Outcome: Number of Days Spent Within Hgb Range ( ±0.5 g/dL and ±1 g/dL ) From Baseline Hgb
Description: Time spent with Hgb within range (where range was defined as +-0.5 g/dL and +-1 g/dL from baseline Hgb ) was analyzed. Baseline value of Hgb was recorded pre-dose on Day 1.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 20 | 19 | 20
Days
  Within +/- 0.5 g/dL: number analyzed (Participants) | 20 | 20 | 18 | 19
  Within +/- 0.5 g/dL | 12.82 [6.98 to 21.85] | 14.34 [4.86 to 25.76] | 24.41 [8.94 to 28.00] | 21.15 [10.50 to 28.00]
  Within +/- 1 g/dL: number analyzed (Participants) | 20 | 20 | 18 | 19
  Within +/- 1 g/dL | 27.71 [19.25 to 28.00] | 20.79 [12.76 to 28.00] | 28.00 [24.77 to 28.00] | 28.00 [23.33 to 28.00]

10. Secondary Outcome: Evaluation of Change From Baseline (Pre-dose on Day 1) in Ferritin Over 4 Weeks
Description: Change from Baseline (pre-dose on Day 1) in ferritin over 4 weeks was analyzed. Change from Baseline is the value at indicated time point minus the Baseline value. Model adjusted mean has been presented as LS mean.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Micrograms per liter
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 19 | 18 | 17 | 19
Micrograms per liter | 76.7 (36.31) | -1.6 (37.41) | -76.7 (38.48) | -38.0 (37.27)

11. Secondary Outcome: Evaluation of Change From Baseline (Pre-dose on Day 1) for Transferrin Over 4 Weeks
Description: Evaluation of change from Baseline for ferritin was performed over 4 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Model adjusted mean has been presented as LS mean.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Grams per liter
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 19 | 18 | 17 | 19
Grams per liter | 0.105 (0.0699) | 0.155 (0.0719) | 0.221 (0.0737) | 0.059 (0.0703)

12. Secondary Outcome: Change From Baseline (Pre-dose on Day 1) for Transferrin Saturation Over 4 Weeks
Description: Transferrin saturation is a medical laboratory test and is the ratio of serum iron and total iron-binding capacity, multiplied by 100 and expressed as a ratio. Evaluation of change from baseline for transferrin saturation was performed up to 4 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline value was recorded pre-dose on Day 1. Model adjusted mean values are presented as LS mean values.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed..
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 18 | 18 | 17 | 19
Ratio | 6.4 (3.33) | 11.7 (3.34) | 1.3 (3.42) | -0.1 (3.24)

13. Secondary Outcome: Change From Baseline (Pre-dose on Day 1) for Total Iron Over 4 Weeks
Description: Evaluation of change from Baseline for total iron was performed over 4 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was recorded pre-dose on Day 1. Adjusted mean was presented as LS mean.
Time Frame: Baseline (pre-dose on Day 1) and at Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Micromoles per Liter
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 19 | 18 | 17 | 19
Micromoles per Liter | 4.3 (1.44) | 6.2 (1.47) | 2.5 (1.51) | 0.3 (1.43)

14. Secondary Outcome: Change From Baseline (Pre-dose on Day 1) in Total Iron Binding Capacity Over 4 Weeks
Description: Evaluation of change from Baseline in total iron binding capacity was performed over 4 weeks. Baseline was recorded pre-dose on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Adjusted means are presented as LS means.
Time Frame: Baseline (pre-dose on Day 1) and Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Micromoles per Liter
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 18 | 18 | 17 | 19
Micromoles per Liter | 3.2 (1.05) | 3.7 (1.06) | 5.2 (1.08) | 1.3 (1.03)

15. Secondary Outcome: Change From Baseline (Pre-dose on Day 1) for Red Blood Cells (RBCs) Over 4 Weeks
Description: Change from Baseline in RBCs was a pharmacodynamic (PD) biomarker. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was recorded pre-dose on Day 1. Change from Baseline (pre-dose on Day 1) in RBCs was calculated over 4 weeks.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter (Giga cells per L)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 20 | 19 | 20
10^12 cells per Liter (Giga cells per L)
  Week 1: number analyzed (Participants) | 19 | 20 | 19 | 18
  Week 1 | -0.04 (0.157) | -0.03 (0.189) | -0.06 (0.184) | 0.02 (0.177)
  Week 2: number analyzed (Participants) | 19 | 20 | 17 | 19
  Week 2 | -0.13 (0.191) | -0.14 (0.243) | -0.05 (0.210) | 0.18 (0.771)
  Week 3: number analyzed (Participants) | 16 | 17 | 17 | 18
  Week 3 | -0.22 (0.248) | -0.19 (0.305) | -0.05 (0.229) | 0.01 (0.256)
  Week 4: number analyzed (Participants) | 18 | 18 | 15 | 19
  Week 4 | -0.29 (0.259) | -0.25 (0.337) | -0.03 (0.198) | -0.03 (0.262)

16. Secondary Outcome: Change From Baseline (Pre-dose on Day 1) for Reticulocytes Over 4 Weeks
Description: Evaluation of change from Baseline for reticulocytes was a PD parameter. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline value was recorded pre-dose on Day 1.
Time Frame: Baseline (pre-dose on Day 1) and up to 4 weeks
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 20 | 19 | 20
Percentage change
  Week 1: number analyzed (Participants) | 19 | 20 | 19 | 16
  Week 1 | -0.42 (0.966) | -0.56 (0.751) | 0.03 (0.681) | -0.08 (0.837)
  Week 2: number analyzed (Participants) | 19 | 20 | 17 | 19
  Week 2 | -0.45 (1.072) | -0.49 (0.613) | -0.08 (0.656) | -0.14 (0.737)
  Week 3: number analyzed (Participants) | 16 | 17 | 17 | 18
  Week 3 | -0.34 (1.114) | -0.27 (0.757) | -0.06 (0.634) | -0.35 (0.782)
  Week 4: number analyzed (Participants) | 18 | 18 | 15 | 19
  Week 4 | -0.36 (1.030) | -0.26 (0.533) | -0.03 (0.703) | -0.29 (0.686)

17. Secondary Outcome: Number of Participants Reaching Hgb Stopping Criteria
Description: Participants were analyzed whether they had any increase or decrease from the Baseline Hgb. Hgb increase based stopping criteria included analysis of Increase or decrease of more than or equal to (>=) 2 g/dL from the Baseline (pre-dose on Day 1) was recorded and also the participants with hemoglobin >=13 g/dL were recorded.
Time Frame: Up to 4 weeks
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 20 | 19 | 20
Participants
  Post Baseline Hgb <8.0 | 1 | 1 | 0 | 0
  >=2g/dL Hgb increase post Baseline | 0 | 1 | 1 | 0
  Post Baseline Hgb >=13.0 | 0 | 0 | 1 | 0

18. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. An SAE is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above. Only on-treatment data has been presented.
Time Frame: Up to 4 weeks
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 21 | 20 | 20
Participants
  Any AE | 9 | 7 | 1 | 6
  Any SAE | 0 | 2 | 0 | 2

19. Secondary Outcome: Number of Participants Discontinuing the Study Treatment Due to AEs
Description: Discontinuation of the study drug could be due to safety-related reasons AE. The AEs responsible included anemia, gastrointestinal hemorrhage, and nausea.
Time Frame: Up to 4 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 21 | 20 | 20
Participants | 1 | 2 | 0 | 0

20. Secondary Outcome: Mean Plasma Concentration of GSK1278863 and GSK1278863 Metabolites Over 4 Weeks
Description: Each of the plasma concentration-time plot contained one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot). Plasma concentrations were analyzed for the study drug (GSK1278863), and its metabolites namely GSK2391220 (M2), GSK2531403 (M3), GSK2487818A (M4), GSK2506102A (M5), GSK2531398 (M6), and GSK2531401A (M13). Pharmacokinetic analysis was done on Weeks (W) 2 and 4 at a fixed timely interval of 5 hours (h) on W2 and every hour on W4. Only the data for last visit for W2 and last visit of W4 has been presented.
Time Frame: Up to 4 weeks
Population: Pharmacokinetic (PK) population included all the participants who received at least one dose of the study drug and from whom at least one sample was withdrawn for PK analysis. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863
Number analyzed (Participants) | 21 | 21 | 21
Nanograms per milliliter (ng/mL)
  GSK1278863, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  GSK1278863, Week 2, 7-11h | 0.2292 (0.40031) | 3.3148 (5.89540) | 5.6170 (15.91725)
  GSK1278863, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  GSK1278863, Week 4, 3h | 3.3113 (3.14336) | 17.9009 (12.89917) | 34.7253 (38.79049)
  M2, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  M2, Week 2, 7-11h | 0.4582 (0.28340) | 1.5468 (1.11679) | 4.3165 (3.03668)
  M2, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  M2, Week 4, 3h | 0.6780 (0.42493) | 2.0382 (1.98534) | 7.4288 (3.64287)
  M3, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  M3, Week 2, 7-11h | 0.6386 (0.35940) | 2.1188 (1.60771) | 5.6935 (3.24262)
  M3, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  M3, Week 4, 3h | 0.7921 (0.42785) | 2.2857 (2.03968) | 8.4582 (3.55548)
  M4, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  M4, Week 2, 7-11h | 0.2156 (0.19430) | 0.8121 (0.69622) | 2.3216 (2.75137)
  M4, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  M4, Week 4, 3h | 0.6016 (0.45551) | 1.8355 (1.89643) | 6.1856 (3.24320)
  M5, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  M5, Week 2, 7-11h | 0.1546 (0.11679) | 0.5511 (0.41077) | 1.4581 (0.71612)
  M5, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  M5, Week 4, 3h | 0.1995 (0.22453) | 0.7132 (1.08288) | 1.9972 (0.71061)
  M6, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  M6, Week 2, 7-11h | 0.1776 (0.12140) | 0.6956 (0.47561) | 1.8957 (1.47442)
  M6, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  M6, Week 4, 3h | 0.3235 (0.27845) | 1.0626 (1.35895) | 3.4569 (1.56093)
  M13, Week 2, 7-11h: number analyzed (Participants) | 19 | 18 | 17
  M13, Week 2, 7-11h | 0.4875 (0.38599) | 1.4014 (1.19096) | 3.9647 (1.86947)
  M13, Week 4, 3h: number analyzed (Participants) | 17 | 17 | 17
  M13, Week 4, 3h | 0.4651 (0.35442) | 1.3623 (1.40324) | 5.3494 (2.60236)

21. Secondary Outcome: Number of Participants With Abnormal Hematology and Clinical Chemistry Parameters of Potential Clinical Concern (PCI)
Description: Participants were analyzed up to 6 weeks for hematological and clinical chemistry parameters of PCI whether they had any higher or lower values than the reference range post screening. Normal alkaline phosphatase (ALP) was 0-46 U/L, aspartate amino transferase (AST) 0-42 U/L, ALP 20-125 U/L, total bilirubin 0-1.3 mg/dL, troponin 0-0.1ng/mL, Hgb 12 - 16 g/dL, platelets 140-450 G/L, creatine phosphokinase 29-168 U/L, creatinine 0.57 - 1.25 mg/dL, Potassium 3.6-5.0 mmol/L, hematocrit 38-45%; however, no participants with abnormal hematology and clinical chemistry parameters were recorded.
Time Frame: Up to 6 weeks (including follow-up)
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 21 | 20 | 20
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Abnormal Vital Signs of PCI
Description: Vital signs include systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR). Three measurements of SBP, DBP and HR were recorded from the participant in a supine position for at least 5 minutes (allowing enough time between measurement to completely deflate and loosen the inflatable cuff). Data has been presented for vital signs with values high and low from the reference range.
Time Frame: Up to 6 weeks
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 21 | 20 | 19 | 20
Participants
  DBP, low | 1 | 2 | 2 | 3
  DBP, high | 2 | 2 | 0 | 2
  SBP, low | 0 | 1 | 0 | 1
  SBP, high | 10 | 9 | 6 | 10
  HR, low | 0 | 0 | 0 | 0
  HR, high | 0 | 0 | 3 | 2

23. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings Over Period
Description: Participants were analyzed for any abnormality in ECG and was categorized as abnormal clinically significant and abnormal and clinically insignificant. The parameters that were analyzed for ECG were atrial fibrillation, Atrial premature complex, Bigeminy, First degree AV block (PR interval > 200 msec), Incomplete right bundle branch block, Junctional rhythm, Junctional tachycardia (heart rate >100 beats/min), Left anterior hemi block (synonymous to left anterior fascicular block), Left atrial abnormality, Left axis deviation (QRS axis more negative than -30 degrees), Left bundle branch block, Left ventricular hypertrophy, Myocardial infarction, anterior, Myocardial infarction, inferior, Non-specific ST-T changes, Normal sinus rhythm, Poor R wave progression, Right atrial abnormality, Right QRS axis deviation, bundle block, ventricular hypertrophy, ST depression or abnormality, AV block, arrhythmia, short PR interval, bradycardia, tachycardia, and T-wave abnormality.
Time Frame: Up to 6 weeks
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
Number analyzed (Participants) | 20 | 20 | 19 | 19
Participants
  Abnormal, clinically significant | 10 | 12 | 8 | 12
  Abnormal, not clinically significant | 5 | 6 | 9 | 6

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: Safety population was used to collect AEs and SAEs.
Groups:
- rhEPO: Eligible participants received oral recombinant human erythropoietin (rhEPO ) or darbepoetin once daily for 4 weeks and were followed-up for 2 weeks
Arm/Group | 0.5 mg GSK1278863 | 2 mg GSK1278863 | 5 mg GSK1278863 | rhEPO
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/21 | 0/20 | 2/20
Other Adverse Events (participants affected / at risk) | 3/21 | 1/21 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5 mg GSK1278863 (N=21) | 2 mg GSK1278863 (N=21) | 5 mg GSK1278863 (N=20) | rhEPO (N=20)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5 mg GSK1278863 (N=21) | 2 mg GSK1278863 (N=21) | 5 mg GSK1278863 (N=20) | rhEPO (N=20)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.